CLINICAL TRIAL: NCT00019227
Title: PHASE I/II STUDY OF TAC-EXPRESSING ADULT T-CELL LEUKEMIA (ATL) WITH YTTRIUM-90 (90Y)-RADIOLABELED HUMANIZED ANTI-TAC AND CALCIUM-DTPA
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065240; NCI-96-C-0147K; NCT00001514 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2003-03

CONDITIONS: Lymphoma; Radiation Toxicity
Keywords: stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; radiation toxicity
MeSH Terms: conditions — Lymphoma; Radiation Injuries; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Pentetic Acid; Daclizumab

INTERVENTIONS:
Drug: pentetic acid calcium
Radiation: yttrium Y 90 daclizumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiolabeled monoclonal antibody plus pentetic acid calcium in patients with leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90 daclizumab (90Y daclizumab) when combined with pentetic acid calcium in adults with Tac-expressing T-cell leukemia.
* Determine the therapeutic efficacy and toxicity of this regimen in these patients.
* Monitor patients treated on this regimen for circulating infused antibody (free and labeled) and for the serum concentration of soluble interleukin-2 receptor.
* Evaluate, in a preliminary manner, the immunogenicity of daclizumab.
* Determine the effect of 90Y daclizumab on various components of the circulating cellular immune system.
* Determine whether there is additional urinary excretion of yttrium Y 90 when compared to that observed previously in patients treated without pentetic acid calcium.

OUTLINE: This is a dose escalation study of yttrium Y 90 daclizumab (90Y daclizumab).

Patients receive 90Y daclizumab IV over 2 hours on day 1 and a fixed dose of pentetic acid calcium IV over 5 hours for 3 days. Treatment repeats every 6 weeks for a maximum of 9 courses in the absence of disease progression or circulating antibodies to humanized anti-Tac.

Cohorts of 3-6 patients receive escalating doses of 90Y daclizumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities. Additional patients are treated at the MTD.

Patients are followed at 4-6 weeks.

PROJECTED ACCRUAL: Up to 15 patients will be accrued for the phase I portion of the study. A total of 30 patients will be accrued for the phase II portion of the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adult T-cell leukemia or lymphoma (ATL) of any stage
* Tac expression of malignant cells confirmed by one of the following:

  * At least 10% of peripheral blood, lymph node, or dermal malignant cells reactive with anti-Tac by immunofluorescent staining
  * Soluble interleukin-2 receptor levels greater than 1,000 U/mL (normal geometric mean = 235; 95% confidence intervals = 112-502 U/mL)
* Measurable disease required

  * More than 10% (i.e., strongly Tac-expressing) abnormal cells in peripheral blood considered measurable disease
* All stages of Tac-expressing adult T-cell leukemia are eligible

  * Smoldering ATL patients are eligible only if the symptoms and sites of involvement by ATL are such that there is a medical indication to treat

    * Smoldering ATL, defined as:

      * Lymphocyte count less than 4,000/mm^3
      * Less than 5% abnormal lymphocytes on morphologic exam of peripheral blood
      * No hypercalcemia
      * Lactate dehydrogenase no greater than 1.5 times normal
      * No lymphadenopathy
      * No involvement of extranodal organs except skin or lung
      * No malignant pleural effusion or ascites
* No symptomatic CNS disease due to ATL

  * Concurrent diagnosis of tropical spastic paraparesis allowed
* No detectable levels (i.e., greater than 250 ng/mL) of antibody to study drug as assessed by ELISA

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Greater than 2 months

Hematopoietic:

* Absolute granulocyte count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL (unless directly due to ATL)
* AST/ALT less than 2.5 times normal

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 35 mL/min

Cardiovascular:

* No clinical cardiac failure

Pulmonary:

* No symptomatic pulmonary dysfunction unless due to underlying malignancy

Other:

* HIV negative
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior cytotoxic chemotherapy

Endocrine therapy

* Concurrent corticosteroids allowed

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-10; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A. Waldmann, MD, Study Chair — NCI - Metabolism Branch;MET
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States